CLINICAL TRIAL: NCT03819946
Title: Oesophageal Protection: a Novel Approach to Improving the Safety of Catheter Ablation for Atrial Fibrillation.
Brief Title: Improving Oesophageal Protection During AF Ablation
Acronym: IMPACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. George's Hospital, London (Other)
Collaborators: Attune Medical (Other)
Responsible Party: Principal Investigator, Dr. Mark M. Gallagher, Clinical Lead for Cardiac Electrophysiology and Principal Investigator, St. George's Hospital, London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRAS253844
Record Dates: First submitted 2019-01-20; First posted 2019-01-29 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Esophageal Diseases
Keywords: Esophageal protection; Ablation-related thermal injury; Catheter ablation for AF; Persistent AF ablation
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial with 1:1 randomization to the study protocol or the control. The study group will have esophageal protection utilising the esophageal cooling device. The control group will have standard esophageal protection, using an esophageal temperature probe.
Who Masked: Outcomes Assessor
Masking Description: The endoscopists performing the follow up endoscopy test will be 'blinded' to the randomization of the trial participant, to minimise bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group- esophgeal cooling (Experimental): In this study arm, the participants will have esophageal protection during their catheter ablation procedure, utilizing the esophageal cooling device (Attune Medical, Chicago, IL). During catheter ablation, the cooling device is set to cooling levels.
  Interventions: Device: esophageal cooling device (Attune Medical, Chicago, IL)
- Control group- esophgeal temperature probe (Active Comparator): In this control group, the participants will have esophageal protection utilizing the standard method in current practice, which is an esophageal temperature probe. If recorded temperatures rise above 38 degrees during ablation, ablation treatment is halted in this region.
  Interventions: Other: Standard esophageal temperature probe

INTERVENTIONS:
Device: esophageal cooling device (Attune Medical, Chicago, IL) — The esophageal cooling device is a silicone soft tubing that is designed to be inserted into the esophagus. It is currently used clinically to provide whole body cooling or temperature control for intensive care patients (in medically induced coma or general anesthesia). The tubing is established but not been used in the clinical setting of catheter ablation for AF (which is performed under general anesthesia). During application of ablation energy to the posterior left atrial wall, the tubing is cooled to medium-low levels (25 degrees) and this is controlled by the operator.
  Arms: Study Group- esophgeal cooling
Other: Standard esophageal temperature probe — If the participant is randomized to the control group, then a standard esophageal protection method will be used during their catheter ablation procedure. This comprises of an esophageal temperature probe, inserted whilst the patient is under general anesthesia. If during application of ablation treatment to the posterior left atrial wall causes the esophageal temperature to rise above 38 degrees the ablation treatment is halted in this region. If ablation treatment is incomplete, re-application can be applied again cautiously if temperatures fall back to 37 degrees. Further temperature rise of over 38 degrees at the same region is a contra-indication to further ablation work here.
  Arms: Control group- esophgeal temperature probe

SUMMARY:
Catheter ablation is an established treatment for atrial fibrillation (AF). For those with the more longstanding form of the condition and are graded as longstanding persistent AF, catheter ablation techniques often involve an extensive ablative protocol. This often includes application of ablation energy to the posterior left atrial wall. The left atrial (LA) wall is only on average 5 millimetres away from the esophageal wall. It has been shown that ablation to the posterior LA wall can cause thermal injury to the esophageal wall. Even those that require pulmonary vein isolation only can be at risk of esophageal injury. This injury can impact on patient symptoms as well as increase the risk of an atrio-esophageal fistula being formed. Esophageal protection methods during catheter ablation for AF in current practice is very limited and investigation towards improved approaches, in the form of a randomized clinical trial is required.

The aim or purpose of this research project is to study the effect of esophageal cooling on the incidence of esophageal thermal injury (endoscopy-graded esophageal epithelial lesions and/or the presence of ablation-related gastroparesis with patient symptoms) compared to controls, after a catheter ablation procedure for the treatment of AF.

DETAILED DESCRIPTION:
Overall design This is a randomized controlled trial with 1:1 randomization to study or control group.

Treatment/intervention plan and rationale AF patients awaiting to have a planned catheter ablation procedure as their treatment will be eligible for this study. If they participate, there is a 1:1 randomization to study or control group.

The study group will have their catheter ablation procedure with utilization of esophageal protection using the cooling tubing device (Attune Medical, Chicago IL). The cooling is controlled by the procedural doctor, with temperatures set in the range of patient safety (for example, cooling at 4 degrees). This device is already in use clinically albeit in a different clinical setting. The device is currently used an intensive care setting to provide whole body cooling. It is designed to be inserted into the esophagus. The temperature control does not allow temperatures to go into the extremes, so preserving patient safety.

The control group will have their catheter ablation procedure using standard esophageal protection methods, which is an esophageal temperature probe, to measure for any temperature changes during application of ablation energy. If measured esophageal temperatures reach beyond 38 degrees then ablation is halted in that area.

Follow up endoscopy assessment After the ablation procedure, a follow up upper GI endoscopy test will be performed to review for any ablation-related thermal injury, by a group of endoscopists who are 'blinded' to the randomization of the participant. The follow up endoscopy test will be confirmed with the participant and the timing of this follow up test is within 1 week of their catheter ablation procedure.

Clinic follow up The clinic follow up will remain exactly the same as standard care but at the first clinic (this is 12 weeks or 3 months from the ablation procedure) we will review or ask about any lingering gastro-esophageal symptoms and record this in a basic questionnaire (the GerdQ questionnaire will be used).

ELIGIBILITY:
Inclusion Criteria:

• Any AF patient planned for a catheter ablation procedure or a left atrial ablation protocol that puts them at risk of surrounding structural trauma, including oesophageal injury.

Exclusion Criteria:

* Patients at the age extremities will not be approached for the study. (Paediatric patients or young adults (<aged 18) or older adults over the age of 85)
* Patients having simple or non-left atrial ablation procedures not needing oesophageal protection.
* Patients at high risk of oesophageal bleeding e.g. oesophageal varices.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
• The incidence of catheter ablation related esophageal injury. | 7 days
  The incidence of catheter ablation related esophageal injury will be assessed by endoscopic examination. Evidence of thermal injury or symptomatic gastroparesis will be recorded. The thermal injury scale is graded 0-6. 6 being the worst score indicating severe esophageal injury. Endoscopic evidence of gastroparesis is dictated by presence of significant food residue despite >6 hours of fasting and must be correlated with new patient symptoms post-ablation.

SECONDARY OUTCOMES:
The incidence of esophageal symptoms after catheter ablation treatment. | 3 months
  During clinic assessment follow up, the participant will fill out a reflux symptoms questionnaire. This is called the GerdQ questionnaire (GerdQ stands for: gastro-esophageal reflux disease questionnaire). This is a scoring system of range 0-18, a score of 18 being the worst symptoms outcome.
• The incidence of major adverse outcomes (MACCE- major adverse cardiovascular cerebrovascular events) will be assessed. | 12 months
  The major adverse events recorded includes the risk of cerebrovascular accident, transient ischaemic attacks (TIA) and myocardial infarction (MI). For each condition in this MACCE category- the recorded response will either be 'yes' or 'no' or 'positive' or 'negative'.
Long-term success rate of the catheter ablation procedure as measured from freedom from the treated arrhythmia (atrial fibrillation/atrial tachycardias). | 12 months
  During clinic follow up, Holter monitors (ambulatory ECG monitors) or implantable loop recorders will monitor for any recurrence of the treated arrhythmia. Any recurrence will be recorded to assess longterm success of the catheter ablation treatment (this is objectively measured at 12 months). The outcome response is recorded as either 'yes' or 'no'.

CONTACTS AND LOCATIONS:
Overall Officials: Mark M Gallagher, MD, Principal Investigator — St. George's Hospital NHS Foundation Trust
Locations (1):
- St.George's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will be anonymised and stored securely in the institutional secured electronic database network. During the study, the data will be available to site sub-investigators only.